CLINICAL TRIAL: NCT04850807
Title: Music & MEmory: A Pragmatic TRial for Nursing Home Residents With ALzheimer's Disease
Brief Title: Music & MEmory: A Pragmatic TRial for Nursing Home Residents With ALzheimer's Disease (METRIcAL)_part2
Acronym: METRIcAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Vincent Mor, Florence Pirce Grant University Professor, Professor of Health Services, Policy and Practice, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R33AG057451_part2; R33AG057451 (NIH)
Record Dates: First submitted 2021-04-16; First posted 2021-04-20 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The investigator's primary outcome (staff report of resident agitated and aggressive behaviors) will be evaluated using a parallel design
Who Masked: Investigator
Masking Description: Principal investigator is blinded to allocation of nursing homes to treatment or control conditions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care for managing agitated and/or aggressive behaviors in the nursing home setting
- Music & Memory (Experimental): Music and Memory is a personalized music program in which nursing home staff provide people with dementia with music playlists tailored to their personal history of music preferences at early signs of agitation
  Interventions: Behavioral: Music & Memory

INTERVENTIONS:
Behavioral: Music & Memory — Music and Memory is a personalized music program in which caregivers (nursing home staff, family, or others) provide people with dementia with music playlists tailored to their personal history of music preferences at times when behaviors are likely
  Arms: Music & Memory

SUMMARY:
The purpose of this trial is to test the effects of a personalized music intervention (Music and Memory, Inc.) on agitated and aggressive behaviors for nursing home residents with dementia.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a parallel, pragmatic, cluster randomized control trial of personalized music (Music and Memory) for nursing home residents with moderate to severe dementia living in 54 nursing homes (27 treatment, 27 control) from 4 nursing home corporations. Music and Memory is a personalized music program that uses portable music players to deliver individualized music to people with dementia at times when agitated behaviors are likely.

**This funding mechanism sponsored two parallel trials with different implementation strategies. In this trial, music is preloaded on personalized music devices to increase nursing use of the music with residents. Details of the first parallel trial conducted under this funding mechanism are registered under "R33AG057451_part1."**

The aims of this study are: 1. To use a train-the-trainer model to implement the intervention with ongoing monitoring of the program's adoption and acceptance by nursing home residents with dementia; 2. To estimate the impact of Music and Memory on agitated and aggressive behaviors; and 3. To examine factors associated with variation in providers' adherence to the implementation of Music and Memory.

ELIGIBILITY:
Inclusion Criteria for Nursing Homes:

* Owned by partnering health care corporations
* Medicare / Medicaid-certified
* Have at least 20 eligible residents

Inclusion Criteria for Residents in Eligible Nursing Homes

* Reside in eligible nursing home for last 90 days
* Have a dementia diagnosis

Exclusion Criteria for Nursing Homes:

* recent situations that may affect implementation (for example, bad state or federal quality assurance surveys, leadership turnover, or other competing demands)
* previous use of Music and Memory

Exclusion Criteria for Residents in Eligible Nursing Homes:

* dislikes music
* completely deaf

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mor, PHD, Principal Investigator — Brown University, School of Public Health
Locations (4):
- United States (4):
  - PruittHealth, Norcross, Georgia
  - Vetter Senior Living, Elkhorn, Nebraska
  - CommuniCare Terrapins Division, Blue Ash, Ohio
  - Good Samaritan Society, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: nursing home
Period: Overall Study
Arm/Group | Usual Care | Music & Memory
Started | 489; 27 nursing home | 501; 27 nursing home
Completed | 419; 27 nursing home | 431; 27 nursing home
Not Completed | 70; 0 nursing home | 70; 0 nursing home
Not completed — Death | 50 | 55
Not completed — Discharged | 17 | 13
Not completed — Incomplete baseline data | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Music & Memory | Total
Number analyzed (Participants) | 419 | 431 | 850
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.6 (12.2) | 78.5 (12.5) | 79.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287 | 276 | 563
  Male | 132 | 155 | 287
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 84 | 106 | 190
  White | 313 | 316 | 629
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 18 | 5 | 23
Region of Enrollment [Number; unit: participants]
  United States | 419 | 431 | 850
Cognitive function [Count of Participants; unit: Participants]
  Cognitively intact | 64 | 53 | 117
  Mildly impaired | 95 | 92 | 187
  Moderately impaired | 220 | 233 | 453
  Severely impaired | 40 | 53 | 93

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Agitated and Aggressive Behaviors (Staff Report)
Description: The tool used to interview staff about resident behaviors is the Cohen-Mansfield Agitation Inventory (CMAI). Research staff interview nursing staff who know the resident well to ask how frequently 29 agitated/aggressive behaviors occurred in the past week. There are seven response choices for each item, anchored from never (1) to several times per hour (7). Total scores on the CMAI range from 29 to 203, with higher scores representing more frequent agitated/aggressive behaviors. The CMAI is administered at baseline and follow-up.
Time Frame: 4-months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Music & Memory | Usual Care
Number analyzed (Participants) | 431 | 419
score on a scale | 44.1 (3.1) | 47.9 (3.1)
Statistical Analysis 1: Comparison: Music & Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; average marginal effect = -0.4, 95% CI 2-sided [-6.9 to 6.0], Standard Error of Mean 3.3; Fixed effect covariates: age, sex, race, activities of daily living score, cognitive function score, psychotic disorder, bipolar disease, depression, anxiety, dementia, alzheimer's diagnosis, antidepressant use, antianxietal use, antipsychotic use, history of heart failure, baseline ARBS (exclusive to CMAI model), baseline CMAI (exclusive to ARBS model), indicator of baseline/follow-up score, treatment group, interaction of treatment group and baseline/follow-up score. Random effects: random intercept for nursing home, random intercept for the interaction of baseline/follow-up measure and nursing home, and random intercept for individual. Imputed Outcomes: 37 Control Follow-Up (Both CMAI and ARBS), 37 Treatment Follow-Up (ABRS), 35 Treatment Follow-Up (CMAI)

2. Secondary Outcome: Frequency of Agitated and Aggressive Behaviors (Administrative Data)
Description: The Aggressive Behavior Scale is a 4 item measure describing the frequency of physical behavioral symptoms directed toward others; verbal behavioral symptoms directed toward others; other behavioral symptoms not directed toward others; and behaviors related to resisting necessary care. For each item, frequency in the past week is reported as: behavior not exhibited (0); behavior occurred 1-3 days (1); behavior occurred 4-6 days (2); or behavior occurred daily (3). The Aggressive Behavior Scale ranges from 0 to 12, with higher scores indicating more frequent agitated and/or aggressive behaviors. Mean total scores will be compared for treatment and control populations.
Time Frame: 4 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Music & Memory | Usual Care
Number analyzed (Participants) | 431 | 419
score on a scale | 0.38 (0.07) | 0.31 (0.07)
Statistical Analysis 1: Comparison: Music & Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; Average Marginal Effect = 0.10, 95% CI 2-sided [-0.06 to 0.26], Standard Error of Mean 0.08; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Antipsychotic Use
Description: Any antipsychotic use in the past week, based on Minimum Data Set (standardized assessment of nursing home residents). Comparison of percent with any use will be compared for treatment and control populations. Measure type of mean is chosen based on adjusted percentage with standard errors from a multilevel, difference in difference regression models.
Time Frame: 4 months
Measure: Mean (Standard Error); unit: adjusted percentage of participants
Arm/Group | Music & Memory | Usual Care
Number analyzed (Participants) | 431 | 419
adjusted percentage of participants | 43.6 (2.3) | 39.7 (2.2)
Statistical Analysis 1: Comparison: Music & Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; average marginal effect = 4.0, 95% CI 2-sided [-2.3 to 10.2], Standard Error of Mean 3.2; Fixed effect covariates: baseline medication use, age, sex, race, activities of daily living score, cognitive function score, psychotic diagnosis, depression, anxiety, dementia, asthma, ARBS score, treatment group. Random effects: random intercept for nursing home Imputed Outcomes: 37 Control Follow-Up , 35 Treatment Follow-Up

4. Secondary Outcome: Antianxietal Use
Description: Any antianxietal use in the past week , based on Minimum Data Set (standardized assessment of nursing home residents). Comparison of adjusted percent with any use will be compared for treatment and control populations. Measure type of mean is chosen based on adjusted percentage with standard errors from a multilevel, difference in difference regression models.
Time Frame: 4 months
Measure: Mean (Standard Error); unit: adjusted percentage of participants
Arm/Group | Music & Memory | Usual Care
Number analyzed (Participants) | 431 | 419
adjusted percentage of participants | 32.3 (2.5) | 33.7 (2.6)
Statistical Analysis 1: Comparison: Music & Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; average marginal effect = -1.4, 95% CI 2-sided [-8.5 to 5.6], Standard Error of Mean 3.6; Results are adjusted for baseline medication use, age, sex, race, activities of daily living score, cognitive function score, psychotic diagnosis, depression, anxiety, dementia, asthma, ARBS score, treatment group. The model includes a random intercept for nursing home

5. Secondary Outcome: Antidepressant Use
Description: Any antidepressant use in the past week, based on Minimum Data Set (standardized assessment of nursing home residents). Comparison of percent with any use will be compared for treatment and control populations. Measure type of mean is chosen based on adjusted percentage with standard errors from a multilevel, difference in difference regression models.
Time Frame: 4 months
Measure: Mean (Standard Error); unit: adjusted percentage of participants
Arm/Group | Music & Memory | Usual Care
Number analyzed (Participants) | 431 | 419
adjusted percentage of participants | 63.8 (1.8) | 68.6 (1.8)
Statistical Analysis 1: Comparison: Music & Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; average marginal effect = -4.8, 95% CI 2-sided [-9.8 to 0.1], Standard Error of Mean 2.5; [other analysis details as in outcome 3, analysis 1]

6. Secondary Outcome: Hypnotic Use
Description: Any hypnotic use in the past week, based on Minimum Data Set (standardized assessment of nursing home residents). Comparison of percent with any use will be compared for treatment and control populations.
Time Frame: 4 months
Measure: Number; unit: unadjusted percentage of participants
Arm/Group | Music & Memory | Usual Care
Number analyzed (Participants) | 431 | 419
unadjusted percentage of participants | 1.62 | 0.95

7. Secondary Outcome: Depression
Description: The Patient Health Questionnaire is a 9-item screening assessment for depression severity. For each item, respondents indicate the frequency of the symptom in the past 2 weeks using the following choices: never or one day (0); 2-6 days (1); 7-11 days (2); or 12-14 days (3). Total scores range from 0 to 27, with higher scores indicating more frequent depressive symptoms. Average total scores will be compared for treatment and control populations.
Time Frame: 4 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Music & Memory | Usual Care
Number analyzed (Participants) | 431 | 419
score on a scale | 2.33 (0.44) | 1.61 (0.47)
Statistical Analysis 1: Comparison: Music & Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; average marginal effect = -0.31, 95% CI 2-sided [-1.03 to 0.41]; Fixed effect covariates: age, sex, race, activities of daily living score, cognitive function score, psychotic disorder, bipolar disease, depression, anxiety, dementia, alzheimer's diagnosis, antidepressant use, antianxietal use, antipsychotic use, history of heart failure, baseline ARBS (exclusive to CMAI/PHQ-9 model), baseline CMAI (exclusive to ARBS/PHQ-9 model), indicator of baseline/follow-up score, treatment group, interaction of treatment group and baseline/follow-up score. Random effects: random intercept for nursing home, random intercept for the interaction of baseline/follow-up measure and nursing home, and random intercept for individual. Imputed Outcomes: 37 Control Follow-Up (Both CMAI and ARBS), 37 Treatment Follow-Up (ABRS), 35 Treatment Follow-Up (CMAI)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during each resident's 4-month follow-up period.
Arm/Group | Usual Care | Music & Memory
All-Cause Mortality (participants affected / at risk) | 50/489 | 55/501
Serious Adverse Events (participants affected / at risk) | 0/489 | 0/501
Other Adverse Events (participants affected / at risk) | 0/489 | 0/501

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT04850807/Prot_SAP_000.pdf